CLINICAL TRIAL: NCT06792747
Title: Evaluation of Diagnostic Accuracy of Artificial Intelligence in Treatment Planning for Non-growing Class II Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Israa Abuobieda Ibrahim Elbagari, Master Degree student at the department of orthodontics, Cairo University
Other Study IDs: AI accuracy for Class II 2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-01

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the diagnostic accuracy of artificial intelligence in non-growing class II cases. The main question it aims to answer is:

Is Artificial Intelligence (AI) accurate in choosing a treatment modality for non-growing class II cases -whether to camouflage or surgical treatment?

participants already undergone orthodontic treatment, their pre-treatment and post-treatment records will be collected from the archive of orthodontic department at Cairo university

ELIGIBILITY:
Inclusion Criteria:

cases of non-growing patients with class II malocclusion

Exclusion Criteria:

Growing patient with class II malocclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian non-growing individuals with class II malocclusion
Sampling Method: Non-Probability Sample
Enrollment: 193 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Artificial intelligence in choosing\predicting the best treatment modality | from enrollment to the end of treatment at 1 year